CLINICAL TRIAL: NCT06142786
Title: Examine the Effectiveness of Individualized Alpha Neurofeedback for Children With ADHD, a Triple-blinded Randomised Control Trial
Brief Title: Individualized Alpha Neurofeedback for ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Winnie Wan Yee Tso (Dr), Clinical Assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADHD_NF_HKU
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: ADHD
Keywords: ADHD; Neurofeedback
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Once eligible participants are enrolled in this study, they will be randomly allocated either to the neurofeedback intervention group or the sham feedback group. Participants in both groups will receive treatment/sham treatment at the same period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, their parents/guardians, the neurofeedback/sham feedback trainer, the investigator, and outcome assessors will be blinded to the allocation of conditions. An independent senior research assistant from our team, who is not involved in the mentioned roles, will execute the random allocation algorithm and set the neurofeedback training protocol (either verum or sham) before each visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individualized alpha neurofeedback (Experimental)
  Interventions: Behavioral: Enhancing the individualized upper alpha frequency band and suppressing the lower alpha band.
- Sham neurofeedback (Sham Comparator)
  Interventions: Behavioral: Sham neurofeedback

INTERVENTIONS:
Behavioral: Enhancing the individualized upper alpha frequency band and suppressing the lower alpha band. — Real time visual feedback will be given the participants, such that as the higher/lower alpha power increases (relative to the mean value in the pre-training resting state EEG recording) a plane on the screen will move horizontally (the movement is correspondent to the magnitude of upper/lower alpha ratio), and the animation will change based on EEG parameter every 2 seconds. EMG-based feedback is also provided, such that if the children's EMG level is too high the plane will drop (vertical movement). Participants are instructed to 'fly' the plane as far as possible.
  Arms: Individualized alpha neurofeedback
Behavioral: Sham neurofeedback — The sham neurofeedback protocol was identical to the verum neurofeedback protocol except that the animation (horizontal plane movement) was based on the EEG results of another participant. EMG-based feedback will still be provided for the sham condition
  Arms: Sham neurofeedback

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is one of the most prevalent neurodevelopmental disorders, characterised by inattention, hyperactivity, and impulsivity. Although pharmacotherapy is considered the first-line treatment for ADHD at all ages (at least for severe cases), non-pharmacological therapies might be equally effective without the risk of drug side effects. Some studies have shown that electroencephalographic (EEG) neurofeedback improves parent-rated ADHD symptoms in children and adolescents. However, whether neurofeedback is an effective treatment for ADHD is still under debate.

Several issues may hinder the evaluation of the effectiveness of neurofeedback treatment in previous studies. Firstly, previous neurofeedback studies did not utilize effective neurophysiological markers for ADHD. Theta/Beta ratio, the most common neurofeedback marker for treating ADHD in the past two decades, has recently been suggested to be only weakly correlated to individuals' attention. Secondly, previous studies mostly used the norm of the EEG markers in age/gender matched healthy children as the training target for ADHD children, which largely ignored the individual variations in EEG acquisition. Third, most of the previous studies lack a rigorous study design, for comparing neurofeedback with a 'placebo' condition and evaluating its specific and non-specific effects.

In the current studies, we propose to conduct a sham-controlled, triple-blind trial to evaluate the effectiveness of an individual-based neurofeedback treatment for ADHD children and adolescents. The EEG marker for neurofeedback in treating ADHD would be the individualized lower/higher alpha band power, based on the recent methodological advances in EEG spectrum processing (1/f model fit and individualized peak alpha frequency modelling) . The training target will be individualized and defined according to the neurophysiological pattern shown in pre-training resting-state conditions, and thus each participant will be trained to achieve their own optimum state of engagement. Sham neurofeedback will be used as a placebo condition, controlling for the non-specific effect of neurofeedback. The study will be triple-blinded (i.e, participants, individuals who administered treatment or intervention, and those who assessed the outcomes were masked).

DETAILED DESCRIPTION:
120 ADHD children will be invited to join the RCT neurofeedback training. They will be randomly assigned to one of two groups (neurofeedback group, sham feedback group, ). For the neurofeedback group participants will undergo an 4-week neurofeedback training (twice a week); for the sham feedback group， participants will undergo an 4-week sham feedback training (twice a week), All the groups will conduct cognitive and EEG tests before and after the 4-week period and the investigators will follow up with all the participants immediately after the training and 6-month after the training. When recruiting, participants and parents of the participants will be notified that their children are likely to be assigned to one of the three groups, and for the neurofeedback and sham feedback group, the parents and participants will not know which condition they are enrolled in, until the end of the study. By the end of the study, participants from the sham feedback group will be given an opportunity to rejoin a neurofeedback session for compensation.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilment of the DSM-IV-TR criteria for ADHD
* No intention to use new medication/change dosage/join new non-pharmacological treatment program during the intervention period.

Exclusion Criteria:

* Diagnosis of cerebral palsy/ history of structural brain abnormalities on CT/ MRI;
* full-scale IQ score (FSIQ) < 70;
* A history of seizure or prior electroencephalogram abnormalities related to epilepsy.
* Having comorbid psychiatric disorders, including schizophrenia or schizoaffective disorder, bipolar disorder, borderline personality disorder, epilepsy, or traumatic brain injury; current substance abuse or dependence
* Planned other behavioural/durg treatment during the intervention period

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Strengths and Weaknesses of Attention-Deficit/Hyperactivity Symptoms and Normal Behavior Scale (SWAN) | prior to the intervention, immediate after the interventions & 6 months after the intervention
  The Chinese SWAN is a validated instrument for the assessment of ADHD symptoms in Chinese children in Hong Kong. The SWAN questionnaire was originally devised by Swanson et al in 2005 based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for ADHD.
Conners CPT (Conners Continuous Performance Test) | prior to the intervention, immediate after the intervention
  The Conners Continuous Performance Test (CPT) is a computerized neuropsychological assessment designed to evaluate attention, impulsivity, and vigilance in children and adolescents aged 8-18 years. The test involves the presentation of letters on a computer screen, where the participant must respond to specific target letters while ignoring others. The Conners CPT provides measures of response time, errors, and variability, which can aid in the identification of attention deficit hyperactivity disorder (ADHD) and other attention-related problems.

SECONDARY OUTCOMES:
PedsQL (Pediatric Quality of Life Inventory) | prior to the intervention, immediate after the intervention & 6 months after the intervention
  The Pediatric Quality of Life Inventory (PedsQL) is a reliable and validated instrument for assessing health-related quality of life in children and adolescents aged 2-18 years. It consists of 23 items, covering four domains: physical functioning, emotional functioning, social functioning, and school functioning. The PedsQL is designed to measure the impact of various health conditions on children's daily lives and well-being.
SDQ (Strengths and Difficulties Questionnaire) | prior to the intervention, immediate after the intervention 6 months after the intervention
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioral screening questionnaire for children and adolescents aged 2-17 years. It consists of 25 items, covering five domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. The SDQ is designed to help identify mental health problems and promote emotional well-being in children and adolescents.
The Child Behavior Checklist (CBCL) | prior to the intervention, immediate after the intervention & 6 months after the intervention
  The CBCL is a 120 item parent-report, which provides a measure of behavioral and emotional functioning and social competence of youth, aged six to 18
the Wechsler Intelligence Scale for Children (WISC): | prior to the intervention, immediate after the intervention
  The Wechsler Intelligence Scale for Children (WISC) is a comprehensive, standardized intelligence test designed for children and adolescents aged 6-16 years. The WISC measures cognitive abilities across various domains, including verbal comprehension, visual-spatial abilities, fluid reasoning, working memory, and processing speed. The test consists of several subtests, each designed to assess different aspects of cognitive functioning. The WISC is widely used in educational and clinical settings to help identify learning difficulties, intellectual giftedness, and other cognitive issues that may impact a child's academic performance and daily functioning

CONTACTS AND LOCATIONS:
Overall Officials: Winnie WY Tso, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Li Ka Shing Faculty of Medicine, Hong Kong, Hong Kong, Hong Kong